CLINICAL TRIAL: NCT00766558
Title: Study of the Efficacy of Written Emotional Disclosure on Eating Disorder Pathology
Brief Title: The Effects of Written Emotional Disclosure on Eating Disorder Pathology in a Clinical Eating Disordered Population
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 28860
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Eating Disorder
Keywords: anorexia; bulimia; eating disorder not otherwise specified
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders; Anorexia; Bulimia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1 Disclosure: Traumatic writing prompts provided. Participant is assigned a potential stress-producing topic for written disclosure.
- 2 control: Received nontraumatic writing prompts. Participant assigned a non-stressful writing condition

SUMMARY:
A technique that has been found to be effective at relieving the physical and psychological symptoms associated with inhibiting emotions and emotional thoughts is written emotional disclosure. The goal of this study is to evaluate the effectiveness of written emotional disclosure on the remediation of eating disorder behaviour, cognitions, and management of emotions.

DETAILED DESCRIPTION:
New Partial program participants complete a packet of questionnaires during their initial appointment, which will be used as baseline levels of eating disorder symptoms and psychological health. Participants will complete the writing as part of their eating disorder therapy. The writing will be completed individually. The writing will consist of continuous writing for fifteen minutes on three consecutive days. The experimental group will write about traumatic or stressful experiences, while the control group will objectively describe events. A post-writing packet of questionnaires will be completed one week after completing the writing. A follow-up evaluation will occur four-weeks after completion of the post-writing packet and will include completing a packet of questionnaires and debriefing.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign consent form

Exclusion Criteria:

* Unwilling to sign consent form

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients in the Penn State Hershey Adolescentand Adult Eating Disorders Partial Hospitalization Program
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Testing and behavioral changes | 6-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Levine, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Pennebaker, J. W., Chung, C. K., Ireland, M., Gonzales, A., and Booth, R. J. (2007). The development and psychometric properties of LIWC2007. Retrieved June 1, 2008, from Linguistic Inquiry and Word Count web site http://www.LIWC.net/liwcdescription.php
- [Background] Pennebaker, J. W. and Francis, M. E. (1996). Cognitive, emotional, and language processes in disclosure. Cognition and Emotion, 10, 601-626.
- [Background] Pennebaker JW, Kiecolt-Glaser JK, Glaser R. Disclosure of traumas and immune function: health implications for psychotherapy. J Consult Clin Psychol. 1988 Apr;56(2):239-45. doi: 10.1037//0022-006x.56.2.239. No abstract available. PMID 3372832
- [Background] Petrie KJ, Booth RJ, Pennebaker JW. The immunological effects of thought suppression. J Pers Soc Psychol. 1998 Nov;75(5):1264-72. doi: 10.1037//0022-3514.75.5.1264. PMID 9866186
- [Background] Petrie KJ, Fontanilla I, Thomas MG, Booth RJ, Pennebaker JW. Effect of written emotional expression on immune function in patients with human immunodeficiency virus infection: a randomized trial. Psychosom Med. 2004 Mar-Apr;66(2):272-5. doi: 10.1097/01.psy.0000116782.49850.d3. PMID 15039514
- [Background] Quinton, S. and Wagner, H. L. (2005). Emotional expression, alexithymia, and characteristics associated with eating psychopathology in non-clinical women. Personality and Individual Differences, 38, 1163-1173.